CLINICAL TRIAL: NCT03494504
Title: A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Phase 3 Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solutions (0.25% and 0.5%) Compared to Vehicle in the Conjunctival Allergen Challenge (Ora-CAC®) Model of Acute Allergic Conjunctivitis
Brief Title: ALLEVIATE Trial - A Phase 3 Trial in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-008
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2018-04

CONDITIONS: Allergic Conjunctivitis
Keywords: reproxalap
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Reproxalap Ophthalmic Solution (0.5%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.5%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered once.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Reproxalap Ophthalmic Solution (0.5%) — Reproxalap Ophthalmic Solution (0.5%) administered once.
  Arms: Reproxalap Ophthalmic Solution (0.5%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered once.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solutions in Subjects with Acute Allergic Conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race
* have a positive history of ocular allergies and a positive skin test reaction to a seasonal allergen (grasses, ragweed, and/or trees) as confirmed by an allergic skin test at the Screening Visit or within the past 24 months;
* have a calculated visual acuity of 0.7 logMAR or better in each eye as measured using an ETDRS chart

Exclusion Criteria:

* have known contraindications or sensitivities to the use of the investigational product or any of its components
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium or a diagnosis of dry eye)
* have had ocular surgical intervention within three (3) months prior to Visit 1 or during the trial and/or a history of refractive surgery six (6) months prior to Visit 1 or have ocular or systemic surgery planned during the study or within 30 days after
* have a known history of retinal detachment, diabetic retinopathy, or active retinal disease
* have the presence of an active ocular infection (bacterial, viral or fungal) or positive history of an ocular herpetic infection at any visit
* be a female who is currently pregnant, planning a pregnancy, lactating, not using a medically acceptable form of birth control throughout the trial duration, or has a positive urine pregnancy test at Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cornea Consultants of Arizon, Phoenix, Arizona
  - Eye Site Sacramento, Sacramento, California
  - East West Eye Institute, Torrance, California
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Andover Eye Associates, Andover, Massachusetts
  - Eye Clinics of South Texas, San Antonio, Texas
  - R & R Research, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reproxalap Ophthalmic Solution (0.25%); Reproxalap Ophthalmic Solution (0.5%): Reproxalap administered once 10 minutes prior to pollen exposure
- Vehicle Ophthalmic Solution: Vehicle administered once 10 minutes prior to pollen exposure
Period: Overall Study
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Started | 109 | 100 | 109
Completed | 109 | 100 | 109
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 109 | 100 | 109 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 90 | 90 | 102 | 282
  >=65 years | 19 | 10 | 7 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 63 | 197
  Male | 37 | 38 | 46 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 9 | 46
  Not Hispanic or Latino | 90 | 82 | 100 | 272
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 9 | 15 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 11 | 19 | 17 | 47
  White | 85 | 71 | 76 | 232
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109 | 100 | 109 | 318
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 1 | 2 | 0 | 3
  Blue | 26 | 25 | 27 | 78
  Brown | 57 | 52 | 64 | 173
  Hazel | 13 | 9 | 10 | 32
  Green | 10 | 11 | 8 | 29
  Gray | 2 | 1 | 0 | 3
  Other | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 1 | 2 | 0 | 3
  Blue | 26 | 25 | 27 | 78
  Brown | 57 | 52 | 64 | 173
  Hazel | 13 | 9 | 10 | 32
  Green | 10 | 11 | 8 | 29
  Gray | 2 | 1 | 0 | 3
  Other | 0 | 0 | 0 | 0
Randomization Stratum [Count of Participants; unit: Participants] — Itching scale is 0 to 4 (0 = none, 4 = severe)
  Participants
    <= 2.7 Average Baseline Itching Score | 41 | 38 | 42 | 121
    > 2.7 and <= 3.5 Average Baseline Itching Score | 31 | 30 | 28 | 89
    > 3.5 Average Baseline Itching Score | 37 | 32 | 39 | 108

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Ocular Itching Score
Description: Subject-reported ocular itching score area under the curve from 10 to 60 minutes post allergen challenge using a 0 to 4 scale (0 = none, 4 = severe) was assessed. The least squares mean was derived from analysis of covariance of area under the curve with baseline as a covariate and treatment as a fixed effect The possible range for area under the curve least squares mean is 0 to 100, where a lower score is better.
Time Frame: Efficacy was assessed after a single dose; baseline was assessed approximately two weeks before dosing.
Population: Intent-to-treat population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale*minutes
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 109 | 100 | 109
units on a scale*minutes | 52.003 (3.3053) | 60.040 (3.4552) | 74.657 (3.3076)

2. Secondary Outcome: Number of Subjects With Two-point Reduction in Itching Score
Description: The number of within subject 2-point responders (2-point reduction in itch score from 20-60 minutes post-challenge) using a 0 to 4 scale (0 = least, 4 = most) from the 5-minute post-challenge itch score at baseline was assessed.
Time Frame: Efficacy was assessed after a single dose; baseline was assessed approximately two weeks before dosing.
Population: Intent-to-treat population with observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 109 | 100 | 109
Participants | 88 | 77 | 77
Statistical Analysis 1: Comparison: Reproxalap Ophthalmic Solution (0.25%); Test type: Superiority; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.46 to 3.84]
Statistical Analysis 2: Comparison: Reproxalap Ophthalmic Solution (0.5%); Test type: Superiority; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.11 to 2.94]

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately two months.
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/100 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/100 | 0/109
Other Adverse Events (participants affected / at risk) | 31/109 | 41/100 | 1/109
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=109) | Reproxalap Ophthalmic Solution (0.5%) (N=100) | Vehicle Ophthalmic Solution (N=109)
General disorders and administration site conditions (General disorders) | 31 | 41 | 1 — Transient and self-limiting instillation site irritation that resolved in all cases. All adverse events were deemed mild in severity by the Principal Investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03494504/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03494504/SAP_001.pdf